CLINICAL TRIAL: NCT04980937
Title: Ski- and Snowboard Related Open Peroneal Nerve Injury: a 20- Year Retrospective Case Series Study
Brief Title: Peroneal Nerve Injury: a 20- Year Retrospective Case Series Study
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: IBK-peroneus_2020
Record Dates: First submitted 2021-04-22; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-04

CONDITIONS: Traumatic Injury; Peroneal Nerve Injury; Sport Injury
Keywords: Ski accident; traumatic; peroneal nerve injury; reconstructive surgery; case series
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with perineal nerve damage after ski injury: Retrospectively aquired patients from insight in medical records. All patients with perineal nerve damage after ski injury in the time period of question were enrolled. Inclusion required operative management of the injury interns of microsurgical reconstruction of peroneal nerve.
  Interventions: Procedure: Microsurgical reconstruction of peroneal nerve with or w/o nerve grafts.

INTERVENTIONS:
Procedure: Microsurgical reconstruction of peroneal nerve with or w/o nerve grafts.

SUMMARY:
In a 20-year retrospective study, all skiers and snowboarders with a peroneal nerve injury at the fibular head treated surgically at the Department of Plastic, Reconstructive and Aesthetic Surgery at the Medical University of Innsbruck, Austria, were included. Covering a period from 1999/2000 to 2018/2019.

DETAILED DESCRIPTION:
All data were gained in a clinical routine context, and the study design was retrospective. The work was approved by the local ethics committee of the Medical University of Innsbruck, Innsbruck, Austria (EK Nr.: 1300/2019). We reviewed medical charts from over a 20-year period, including all patients with a PNI after a ski- or snowboard-related accident requiring surgical intervention at the Department of Plastic, Reconstructive and Aesthetic Surgery of the Medical University of Innsbruck, Austria.

We analyzed the demographical data, including age, gender, and citizenship, as well as included variables concerning the winter sport activity (i.e., ski or snowboard, owned or rented, self-inflicted without collision or collision caused by another skier or snowboarder, professional or recreational athlete). We also analyzed the injury itself (i.e., PNI as main injury, open or closed, motoric, sensible or both, fracture, muscle injury, complete or incomplete transection), as well as the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Skiers and snowboarders
* treated with a peroneal nerve injury at the fibular head
* time frame January 1999 to Dicember 2019

Exclusion Criteria:

* Different injury mechanism
* injury of a different nerve than peroneal nerve

Ages: 10 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients who suffered a peroneal nerve injury caused by the sharp edge of a ski or snowboard and required surgical intervention.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 1999-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Successful nerve reconstruction | 1 year
  Functional reconstruction (Janda degree >3; 2-point discrimination)

IPD SHARING:
Plan to Share IPD: No